CLINICAL TRIAL: NCT06548464
Title: Development and Validation of Interpretable Machine Learning Models for Prognosis in Gastric Cancer Patients: a Multicenter Retrospective Study
Brief Title: Interpretable Machine Learning Models for Prognosis in Gastric Cancer Patients
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2024KY154
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stomach Neoplasms; Gastrectomy; Machine Learning
Keywords: Machine Learning; Prognosis; Stomach Neoplasms; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter, retrospective cohort study aimed to develop and validate an explainable prediction model for prognosis after gastrectomy in patients with gastric cancer.

DETAILED DESCRIPTION:
This multicenter, retrospective cohort study aimed to develop and validate an explainable prediction model for prognosis after gastrectomy in patients with gastric cancer. The study included patients who underwent radical gastrectomy for primary gastric or gastroesophageal junction cancer across multiple institutions in China.

The primary objective was to create a machine learning-based model to predict postoperative outcomes following gastrectomy, using readily available clinical and pathological parameters. The main outcome of interest was early recurrence within 2 years after surgery, which significantly impacts overall prognosis.

The study employed various machine learning algorithms to develop prediction models, which were then compared and validated. Model performance was assessed through measures such as area under the receiver operating characteristic curve (AUC), calibration, and Brier score. The SHapley Additive exPlanations (SHAP) method was used to interpret the model and rank feature importance.

This research aims to provide clinicians with a tool for identifying patients at higher risk of poor postoperative outcomes who may benefit from more intensive post-operative monitoring and early intervention strategies, potentially improving prognosis for gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary gastric or gastroesophageal junction cancer
* Underwent radical gastrectomy
* Complete clinical and pathological data available

Exclusion Criteria:

* Presence of distant metastases before surgery
* Non-adenocarcinoma histology
* Incomplete follow-up data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes adult patients of all genders who were diagnosed with primary gastric or gastroesophageal junction adenocarcinoma and underwent radical gastrectomy at participating institutions in China. The study population represents a diverse group of gastric cancer patients, varying in age, tumor stage, and treatment approaches, including those who received neoadjuvant therapy. This cohort aims to provide a comprehensive representation of gastric cancer patients treated with curative intent, allowing for the development and validation of prognostic models applicable to a wide range of clinical scenarios.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Survival | Up to 5 years after surgery
  Assessment of overall survival outcomes in gastric cancer patients after gastrectomy.

SECONDARY OUTCOMES:
Early Recurrence | Within 2 years after surgery
  Incidence of cancer recurrence within 2 years after gastrectomy.
Late Recurrence | From 2 years up to 5 years after surgery
  Incidence of cancer recurrence occurring more than 2 years after gastrectomy.
Postoperative Complications | Within 30 days after surgery
  Incidence and severity of complications following gastrectomy.
Neoadjuvant Treatment Efficacy | From initiation of neoadjuvant therapy to surgery (typically 2-3 months)
  Assessment of tumor response to neoadjuvant therapy before gastrectomy.
5-Year Survival Rate | 5 years after surgery
  Percentage of patients alive 5 years after gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Chang-ming Huang, Fuzhou, Fujian, China